CLINICAL TRIAL: NCT03439683
Title: Knowledge, Attitudes And Practices Among Critical Care Professionals Towards Patient-Ventilator Asynchrony
Brief Title: KAP Asynchrony Survey
Acronym: KAPA
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 61472716.1.0000.0068
Record Dates: First submitted 2018-01-30; First posted 2018-02-20 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Insufficiency; Ventilation Therapy; Complications; Ventilators, Mechanical; Respiration, Artificial
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Physicians: Definition: Physicians working in the ICU for at least 50% of their time in the hospital
  Intervention: Survey about patient-ventilator asynchrony
  Interventions: Other: Survey about patient-ventilator asynchrony
- Nurses: Definition: Nurses working in the ICU for at least 20 hours/week
  Intervention: Survey about patient-ventilator asynchrony
  Interventions: Other: Survey about patient-ventilator asynchrony
- Respiratory Therapists: Definition: Respiratory Therapists working in the ICU for at least 20 hours/week
  Intervention: Survey about patient-ventilator asynchrony
  Interventions: Other: Survey about patient-ventilator asynchrony

INTERVENTIONS:
Other: Survey about patient-ventilator asynchrony — Participants will fill an online survey that asks multiple-choice questions related to knowledge, attitudes and practice related to patient-ventilator asynchrony and also have images of ventilator waveforms wth asynchrony, where they need to identify the type of asynchrony

SUMMARY:
The investigators developed a web-based survey to assess knowledge, attitudes and practice of health care professionals about patient-ventilator asynchrony.

DETAILED DESCRIPTION:
The investigators developed a survey, consisting of 25 multiple choice questions, and including snapshots of mechanical ventilator waveforms to assess the knowledge, attitudes and practice of physicians, nurses and respiratory therapists working in the ICU and caring for patients under mechanical ventilator about patient-ventilator asynchrony. The survey is web-based and will be sent for health professionals working in the ICU of the participating centers. All data will be treated anonymously with the intent of identifying knowledge gaps and inadequate practice that could be remediated by continuous medical education initiatives

ELIGIBILITY:
Inclusion Criteria:

* current working in the ICU as a physician, nurse or respiratory therapist

Exclusion Criteria:

* refusal to sign informed consent
* incomplete survey (less than 80% of the questions answered)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: health professionals working in the ICU of participating hospitals, involved with patient care.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-03-26 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Survey score | in 30 minutes (at survey completion)
  the number of correct answers given to knowledge part of the survey

SECONDARY OUTCOMES:
attitudes score | in 30 minutes (at survey completion)
  the number of desirable answers given to attitudes part of the survey
Practice score | in 30 minutes (at survey completion)
  the number of desirable answers given to practice part of the survey

CONTACTS AND LOCATIONS:
Overall Officials: Juliana C Ferreira, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas -HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided